CLINICAL TRIAL: NCT07138547
Title: GSL Synthetase Inhibitor Eliglustat Combined With CD30 Target Immunotherapy for the Treatment of of CD30+ Lymphoma: an Open-Label, Randomized, Phase I/II Study
Brief Title: GSL Synthetase Inhibitor Eliglustat Combined With CD30 Target Immunotherapy for the Treatment of of CD30+ Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-097
Record Dates: First submitted 2025-08-14; First posted 2025-08-24 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — eliglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with CD30+ lymphoma (Experimental): Eliglustat 63mg will be administered twice daily in patients who are CYP2D6 extensive metabolizers (EMs), or intermediate metabolizers (IMs), in the first 14 days and the following every other week until 24 weeks. For patients who still benefit from the trial, eliglustat 63mg will be administered twice daily every other week to 96 weeks.
  CD30 target immunotherapy: Brentuximab Vedotin 1.2-1.8mg/kg day 1 Q21d; or CD30-targeting CAR-T Cell Therapy( Application should be in accordance with the specific instructions for each cell preparation).
  Interventions: Drug: Eliglustat, CD30 target immunotherapy

INTERVENTIONS:
Drug: Eliglustat, CD30 target immunotherapy — Eliglustat 63mg will be administered twice daily in the first 14 days and the following every other week.
  CD30 target immunotherapy：Brentuximab Vedotin or CD30-targeting CAR-T Cell Therapy.

SUMMARY:
Targeted therapy against the CD30 molecule has achieved some progress in CD30-positive Hodgkin lymphoma, but its efficacy remains unsatisfactory. Previous studies have demonstrated that N-glycan modifications in the extracellular domain of target proteins can disrupt immune synapse formation with CAR-T cells. Our preliminary research has shown that ablation of N-glycans on CD30 enhances the anti-tumor effect of CD30-targeted therapy.It is hypothesized that Eliglustat, by inhibiting GSL synthesis,may potentiate the anti-tumor effect. Consequently,we designed and initiated a single-center, open-label phase I/II clinical study to evaluate the efficacy and feasibility of Eliglustat combined with CD30 targeted immunotherapy in patients with CD30-positive lymphoma. The primary endpoint of this study is the safety and efficacy of Eliglustat combined with CD30 targeted therapies.

DETAILED DESCRIPTION:
CD30-targeted therapies, including Brentuximab Vedotin (BV) and CD30-targeted CAR-T cells, have demonstrated limited efficacy in Hodgkin lymphoma,facing challenges such as the lack of durable responses with BV and low complete response (CR) rates with CD30 CAR-T cells. Existing research indicates that N-glycan modifications in the extracellular domain of target proteins may mediate resistance of tumor cells to CAR-T cell therapy.Our preliminary studies have demonstrated that disrupting the CD30 N-glycans in HL tumor cells enhances the anti-tumor effect of CD30-targeted therapy. Based on this, we hypothesize that the glucosylceramide synthase (GSL synthesis) inhibitor Eliglustat, by inhibiting GSL synthesis, may affect N-glycan structure of target proteins and consequently enhancing anti-tumor efficacy.

To further validate the role of Eliglustat in modulating anti-tumor therapy for CD30-positive lymphoma, we designed and initiated a single-center, open label phase I/II clinical study. This study aims to evaluate the efficacy and feasibility of Eliglustat combined with CD30 immunotherapy in patients with CD30-positive lymphoma.Primary Endpoints:1）safety and of Eliglustat combined with CD30 targeted therapies；2）CR rate (%) in the CAR-T cell plus Eliglustat treatment group; Progression-free survival (PFS) in the BV plus Eliglustat treatment group.Secondary Endpoints: 1)Other efficacy indicators (e.g., Objective Response Rate [ORR]) of Eliglustat combined with CD30- targeted molecular therapy; 2) Efficacy biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 75 years of age.
* ECOG performance of less than 2.
* Subjects must have histological confirmation CD30+ lymphoma.
* Patients must have at least one line of antitumor therapy
* Life expectancy of at least 3 months.
* Subjects with lymphoma must have at least one measureable lesion >1cm as defined by lymphoma response criteria.
* Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study, and subjects have recovered to ≤ grade 1 toxicity.
* Subjects with autologous hematopoietic stem-cell transplantation are eligible which must be more than 3 months.
* Subjects must have adequate marrow, live, renal and heart functions.

Exclusion Criteria:

* Participants with CD30- lymphoma.
* CYP2D6 ultra-rapid metabolizers (URMs).
* The patients is taking a CYP2D6 inhibitor and/or concomitantly with a strong or moderate CYP3A inhibitor.
* Subjects with a history of severe hypersensitivity reactions to CD30 target immunotherapy.
* History of allergy or intolerance to study drug components.
* Known brain metastases or active central nervous system (CNS). Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
* Uncontrolled intercurrent illness, including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia) or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
* Known positive test result for human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS).
* Previous or concurrent cancer within 3 years prior to treatment start except for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
* Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered.
* Vaccination within 30 days of study enrollment.
* Active alimentary tract hemorrhage or history of alimentary tract hemorrhage in 1 month.
* Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before the enrollment, and a negative result must be documented
* Being participating any other trials or withdraw within 4 weeks.
* Unable to swallow and retain oral medication, malabsorption syndrome, conditions that significantly impair gastrointestinal function, total gastrectomy or small bowel resection, ulcerative colitis, symptomatic inflammatory bowel disease, partial or complete intestinal obstruction.
* Researchers believe that other reasons are not suitable for clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-26 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects with treatment-related adverse events (AEs) | Up to 120 days after the last dose of study drugs]
  Incidence, nature, and severity of adverse events graded according to the NCI CTCAE v5.0.
CR rate (CRR) in the CAR-T cell plus Eliglustat treatment group | 12 months
  The Complete Response Rate (CRR), as assessed by the investigator, is the proportion of all evaluable subjects who achieve a complete response.
Progression-free survival (PFS) in the BV plus Eliglustat treatment group. | 2 years
  Time from the date of first administration of the study drug to disease progression or death from any cause (any earliest date).

SECONDARY OUTCOMES:
Objective Response Rate [ORR] | 12 months
  The percentage of patients with CR or PR was determined according to the revised lymphoma efficacy evaluation criteria.
CR rate (CRR) /Progression-free survival (PFS)based on CD30 expression level in tumor tissue. | 12 months
  CD30 expression will be evaluated by immunohistochemistry (IHC), and its expression levels will be analyzed for association with CRR/PFS.

CONTACTS AND LOCATIONS:
Locations (1):
- People's Liberation Army General Hospital, Beijing, Beijing Municipality, China